CLINICAL TRIAL: NCT00264914
Title: An Open-Label, Multicenter Study Evaluating the Long-Term Safety and Efficacy of SR121463B in Patients With Syndrome of Inappropriate Antidiuretic Hormone Secretion
Brief Title: Safety and Efficacy of SR121463B in Patients With Syndrome of Inappropriate Antidiuretic Hormone Secretion
Acronym: SIADH Safety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFY5904; LTS10208; EudraCT : 2004-005239-35
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Inappropriate ADH Syndrome; Hyponatremia
Keywords: Inappropriate ADH Syndrome; Hyponatremia
MeSH Terms: conditions — Inappropriate ADH Syndrome; Hyponatremia | interventions — satavaptan

INTERVENTIONS:
Drug: SR121463B

SUMMARY:
To determine the long-term safety and tolerability of SR121463B in patients with syndrome of inappropriate antidiuretic secretion (SIADH). To assess the long-term efficacy of SR121463B in maintaining normal levels of serum sodium in patients with SIADH.

Long term safety is evaluated further in an open label extension study with flexible doses of satavaptan.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years and higher.
* SIADH (the diagnosis of SIADH is based on several criteria including true serum hypoosmolality, inappropriate urinary osmolality, clinical euvolemia, elevated urinary sodium excretion while on normal salt and water intake, and normal renal, adrenal, and thyroid functions: drug induced SIADH will be limited to carbamazepine or derivatives and antidepressants in patients in whom these drugs cannot be discontinued or easily replaced by other drugs)
* Serum sodium between 115 and 132 mmol/L (at least two consecutive serum sodium levels of at least 24 hours apart, from Day -6 to Day -1); for sodium levels between 125 and 132 mmol/L, the spontaneous serum sodium increase between the two assessments on Day -1 should be < 4 mmol/L
* Urinary osmolality >200mOsm/kg H2O
* Urinary sodium > 30 mmol/L

Exclusion Criteria:

* Patients with acute postoperative SIADH
* Presence of dilutional hyponatremia in hypervolemic states such as congestive heart failure and liver disease with ascites
* Presence of signs of hypovolemia (e.g., orthostatic hypotension, increased serum urea nitrogen, increased serum albumin, increased hematocrit, …)
* Administration of other V2 receptor antagonists or demeclocycline or lithium within one month, thiazides diuretics or spironolactone within 15 days, and urea or loop diuretics within two days prior to study drug administration
* Patients with known treated or untreated adrenal deficiency
* Presence of untreated hypothyroidism
* Presence of uncontrolled diabetes with fasting glycemia > 200 mg/dL (> 11.09 mmol/L)
* Presence of clinical and/or electrocardiographical signs of acute myocardial infarction or acute ischemia, or any other clinically significant abnormality according to the Investigator on a 12 lead ECG recording
* Administration of inducers of CYP3A4 (phenytoin, rifampin, Saint John's Wort) or potent and moderate inhibitor so CYP3A4within two weeks prior to study drug administration
* Inadequate hematological, renal and hepatic functions; hemoglobin (Hb) < 9 g/dL, neutrophils < 1,500/mm3, platelets <100,00/mm3, serum creatine >175 µmol/L (or clearance of creatine <30mL/min for where Ethics Committees require this parameter), ALT and /or AST >2x upper limit of normal
* QTcB > 500 ms
* Serum potassium > 5 mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2005-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety : Physical examination, vital signs, adverse events, electrocardiogram, hematology, serum chemistry

SECONDARY OUTCOMES:
Serum sodium

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (11):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- sanofi-aventis Canada, Laval, Canada
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Causeway Bay, Hong Kong
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Geneva, Switzerland

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com